CLINICAL TRIAL: NCT04619498
Title: PediAppRREST - Effectiveness of an Interactive Cognitive Support Tablet App in Reducing Deviations From Guidelines in the Management of Pediatric Cardiac Arrest: a Simulation-based Randomized Controlled Trial
Brief Title: Effectiveness of an Interactive Cognitive Support Tablet App to Improve the Management of Pediatric Cardiac Arrest
Acronym: PediAppRREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Florence (Other); Catholic University of the Sacred Heart (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Silvia Bressan, Assistant professor, Attending Physician in Pediatric Emergency Medicine, MD, PhD., University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIRD191291
Record Dates: First submitted 2020-10-14; First posted 2020-11-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; resuscitation; cognitive aid; mobile app; emergency medicine; simulation; pediatrics
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, three-parallel arm study
Masking Description: Due to the nature of this study, blinding of the participants, investigators and outcome assessors will not be possible. However, data analyses will be performed by a statistician who will be blinded to the allocation arm (PediAppRREST tablet app, PALS pocket reference card, no cognitive aid).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PediAppRREST app (Experimental): The teams assigned to the PediAppRREST arm will manage the simulated scenario of pediatric cardiac arrest using the new PediAppRREST tablet app as a cognitive aid.
  Interventions: Device: PediAppRREST
- CtrlPALS+ (Active Comparator): The teams assigned to the CtrlPALS+ arm will manage the simulated scenario of pediatric cardiac arrest using the American Heart Association Pediatric Advanced Life Support (AHA-PALS) pocket reference card.
  Interventions: Other: AHA-PALS pocket reference card
- CtrlPALS- (No Intervention): The teams assigned to the CtrlPALS- arm will manage the simulated scenario of pediatric cardiac arrest using no PALS-related cognitive aids.

INTERVENTIONS:
Device: PediAppRREST — PediAppRREST is a new audiovisual interactive app for tablets developed to support the management of pediatric cardiac arrest. It sequentially displays directions on recommended management interventions. It was specifically designed to guide the team leader to perform resuscitation interventions in the sequence/timing and modality reported by the American Heart Association Pediatric Advanced Life Support (AHA-PALS) guidelines.
  Arms: PediAppRREST app
Other: AHA-PALS pocket reference card — It is a 10 cm x 16.5 cm, full-color, 2-sided, 6-panel card that shows the American Heart Association Pediatric Advanced Life Support (AHA-PALS) treatment algorithms. By providing a quick reference tool, it serves as a cognitive aid for healthcare providers who either direct or participate in the management of pediatric respiratory and/or cardiovascular emergencies, including cardiac arrest.
  Arms: CtrlPALS+

SUMMARY:
Pediatric cardiac arrest (PCA) has a high mortality and morbidity. Its management is complex and often deviates from guideline recommendations leading to patients' worse clinical outcomes. A new tablet app, named PediAppRREST has been developed by our research group to support the management of PCA. The aim of the study is to evaluate the impact of the PediAppRREST app on the management of a PCA simulated scenario. The investigators have planned to conduct a multicenter, simulation-based, randomized control trial assessing the number of deviations (errors and delays) from international recommendations in PCA management. The hypothesis is that teams who use the PediAppRREST app as a cognitive aid will show fewer deviations from guidelines than teams who use a static paper-based cognitive aid (American Heart Association Pediatric Advanced Life Support pocket reference card) or no cognitive aid, during the management of a simulated PCA scenario.

DETAILED DESCRIPTION:
AIMS

The primary aim of the study is to evaluate the effectiveness of a new tablet app, named PediAppRREST, in reducing deviations from guideline recommendations during pediatric cardiac arrest management.

The secondary aim is to assess the impact of the use of the app on performance and time to accomplish critical interventions for resuscitation, team leader's workload, cardiopulmonary resuscitation quality metrics and overall resuscitation team performance. Furthermore, the study will have the purpose to evaluate the usability of the app.

METHODS

PARTICIPANTS

Participants will be residents in Pediatrics, Emergency Medicine, and Anesthesiology-Intensive Care programs at four Italian University Hospitals (Padova, Firenze, Novara, and Roma). In order to be included in the study, residents must be BLS (Basic Life Support) or P-BLS (Pediatric-Basic Life Support) or PALS (Pediatric Advanced Life Support) or ALS (Advanced Life Support) or ACLS (Advanced Cardiac Life Support) certified, following the American Heart Association (AHA) or the European Resuscitation Council (ERC) recommendations. Additionally, to be eligible for the role of team leader residents must be PALS-certified according to AHA or ERC guidelines. Those residents who are unable to attend the simulation sessions because of maternity/paternity leave, personal/sick leave or training abroad, or who have participated in previous studies using the PediAppRREST app will not be eligible to participate in the trial.

STUDY DESIGN

This will be a multicenter, randomized controlled, three-parallel arm study, conducted in the setting of simulation. All teams, each consisting of three participants, will manage the same scenario of non-shockable pediatric cardiac arrest with the help of one confederate nurse who will act according to a script. Participants will be randomized to teams, and teams to interventions, using a 1:1:1 ratio. According to the allocation into one of three study arms, teams will use, or not use, a different PALS-related cognitive aid during the management of the scenario: 1) an intervention group using the tablet app PediAppRREST; or 2) a control group (CtrlPALS+) using the AHA-PALS pocket reference card; or 3) a control group (CtrlPALS-) not allowed to use any cognitive aid.

All the simulation scenarios will be video recorded, and two independent, previously trained reviewers will report actions performed by the teams and time to accomplish them. Outcomes will be subsequently assessed by two independent outcome assessors using data extracted by video reviewers.

OUTCOMES

The primary outcome of the study will be the number of deviations from AHA PALS guidelines recommendations during the management of pediatric cardiac arrest, defined as delays and errors according to a novel checklist, named c-DEV15plus, based on previously published guidelines, checklists and scoring systems/evaluation tools.

The secondary outcomes will be the performance of critical actions for resuscitation and the time to perform them, the usability of the app (measured by open-ended questions and one validated questionnaire: the System Usability Scale), the team leaders' workload (measured by the validated NASA-Task Load Index), the quality metrics of cardiopulmonary resuscitation (extracted by the manikin's software SkillReporter, Laerdal™) according to AHA guidelines, and the overall team resuscitation performance (measured by the validated Clinical Performance Tool).

SAMPLE SIZE CALCULATION

The investigators calculated the sample size on the basis of the results obtained during two previous studies: one observational simulation-based study and one pilot study conducted to test the app usability. Based on the preliminary results from these studies, using a single factor ANOVA model, 29 scenarios per each of the three groups (PediAppRREST, CtrlPALS+, CtrlPALS-) are necessary to detect a difference of at least 3.00 points on the c-DEV15plus scale using the Tukey-Kramer (Pairwise) multiple comparison procedure at a 5% significance level and 80% power. In consideration that some possible technical problems with video-recording or other study procedures could occur, the investigators aim to increase the recruitment of participating teams by 20% per arm, to compensate for loss of statistical power due to a potential insufficient sample size. Hence, the investigators plan to have 35 scenarios per arm, for a total of 105 scenarios, which will include overall 315 residents who will be divided in teams of three.

STATISTICAL ANALYSIS

The c-DEV15plus scale, the performance and time to accomplish specific resuscitation interventions, workload, overall team performance and cardiopulmonary resuscitation metrics will be compared between groups with one-way ANOVA model, followed by the Tukey-Kramer multiple comparisons adjustment procedure in case of statistical significance. The outcomes will also be analyzed with a linear mixed model considering the team as a cluster to evaluate the influence of participants' characteristics on the outcome. To take into account the correlation of the observations within a team, the investigators will specify an undetermined correlation matrix. In case of a not normal distribution of the model residuals, the investigators will proceed with a transformation in order to normalize the distribution.

CONFIDENTIALITY AND PRIVACY PROTECTION

A written informed consent to take part into the study will be obtained from each participant. To ensure that the data collected remains confidential, all data and videos will be stored on password protected and secured hard-disk drives, that will be stored in locked filing cabinets located at the Department of Women's and Children's health, University of Padova, Italy.

ELIGIBILITY:
Inclusion Criteria:

* to be attending a medical residency training program in Pediatrics, Anesthesiology-Intensive Care or Emergency Medicine
* to be BLS (Basic Life Support) or P-BLS (Pediatric-Basic Life Support) or PALS (Pediatric Advanced Life Suport) or ALS (Advanced Life Support) or ACLS (Advanced Cardiac Life Support) certified, following the American Heart Association (AHA) or the European Resuscitation Council (ERC) courses
* to give consent to participate to the study and to be video-recorded.

Additionally, to be eligible for the role of team leader, residents must be PALS-certified according to AHA or ERC guidelines

Exclusion Criteria:

* to be unable to attend the simulation sessions because of personal leave, maternity/paternity leave, sick leave or training abroad
* participation in previous studies using the PediAppRREST app

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Deviations from American Heart Association Pediatric Advanced Life Support (AHA-PALS) guidelines | Scenario will be video recorded and evaluated by two independent video reviewers. Outcome assessors will score teams' performance by means of the c-DEV15plus score using data extracted by video reviewers through study completion, an average of 15 months.
  Deviations from AHA-PALS guidelines recommendations are defined as delays and errors according to a novel checklist we derived from a previously published checklist, denominated c-DEV (circulation-deviations), published by Wolfe et al. (2020), by integrating it with evidence-based guidelines, previously reported scoring tools and checklists. We named our new modified checklist c-DEV15plus (circulation-deviations 15 plus). It includes 15 items, which represent correct critical actions for pediatric resuscitation. Each item of the c-DEV15plus is scored either as 0, when the action is performed correctly and timely, as described in the item, or as 1, when the action is not undertaken, undertaken incorrectly, or with wrong timing. The sum of the points attributed to the items represents the c-DEV15plus total score, hence ranging from a minimum of 0 to a maximum of 15, with higher scores corresponding to a higher number of deviations from the guidelines and a worse performance.

SECONDARY OUTCOMES:
Recognition of cardiac arrest (pulsenessness) | Scenario will be video recorded and successively two independent video reviewers will assess the pulsessness recognition, through study completion, an average of 15 months.
  The percentage of teams that recognize cardiac arrest (pulselessness).
Time to cardiac arrest (pulsenessness) recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to pulselessness recognition, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the recognition of cardiac arrest (pulselessness), in seconds.
Performance of chest compressions | Scenario will be video recorded and successively two independent video reviewers will assess the performance of chest compressions, through study completion, an average of 15 months.
  Percentage of teams that start chest compressions.
Time to start chest compressions from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to start chest compressions, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the start of chest compressions, in seconds.
Time to start chest compressions from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to start chest compressions, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the start of chest compressions, in seconds.
Performance of ventilation | Scenario will be video recorded and successively two independent video reviewers will assess the start of ventilation, through study completion, an average of 15 months.
  Percentage of teams that start ventilation.
Time to start of ventilation from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to start ventilation, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the start ventilation, in seconds.
Time to start of ventilation from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to start ventilation, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the start ventilation, in seconds.
Use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin | Scenario will be video recorded and successively two independent video reviewers will assess the use of a cardiopulmonary resuscitation board or a rigid surface underneath the manikin, through study completion, an average of 15 months.
  Percentage of teams that use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin.
Time to use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the use of a cardiopulmonary resuscitation board or a rigid surface underneath the manikin, in seconds.
Time to use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to use a cardiopulmonary resuscitation board or a rigid surface underneath the manikin, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the use of a cardiopulmonary resuscitation board or a rigid surface underneath the manikin, in seconds.
Call for emergency team help | Scenario will be video recorded and successively two independent video reviewers will assess the call for emergency team help, through study completion, an average of 15 months.
  Percentage of teams that call for emergency team help.
Time to call for emergency team help from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to call for emergency team help, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to call for emergency team help, in seconds.
Time to call for emergency team help from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to call for emergency team help, through study completion, an average of 15 months.
  Time from the beginning of the scenario to call for emergency team help, in seconds.
Use of electrocardiogram monitoring | Scenario will be video recorded and successively two independent video reviewers will assess the use of electrocardiogram monitoring, through study completion, an average of 15 months.
  Percentage of teams that use of electrocardiogram monitoring.
Time to start electrocardiogram monitoring from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to start electrocardiogram monitoring, through study completion, an average of 15 months.
  Time from cardiac arrest recognition to start of electrocardiogram monitoring, in seconds.
Time to start electrocardiogram monitoring from the beginning of scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to start electrocardiogram monitoring, through study completion, an average of 15 months.
  Time from the beginning of the scenario to start of electrocardiogram monitoring, in seconds.
Administration of a correct first epinephrine | Scenario will be video recorded and successively two independent video reviewers will assess the correct administration of the first epinephrine, through study completion, an average of 15 months.
  Percentage of teams that perform a correct first epinephrine administration (correct dose, dilution, route, followed by a normal saline flush).
Time to first epinephrine administration from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to the first epinephrine administration, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the first epinephrine administration, in seconds.
Time to first epinephrine administration from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to the first epinephrine administration, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the first epinephrine administration, in seconds.
Administration of a correct second epinephrine | Scenario will be video recorded and successively two independent video reviewers will assess the correct administration of the second epinephrine dose, through study completion, an average of 15 months.
  Percentage of teams that perform a correct second epinephrine administration (correct dose, dilution, route, followed by a normal saline flush).
Time to second epinephrine administration from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to second epinephrine administration, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the second epinephrine administration, in seconds.
Time to second epinephrine administration from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to second epinephrine administration, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the second epinephrine administration, in seconds.
Treatment of reversible causes | Scenario will be video recorded and successively two independent video reviewers will assess the correct treatment of reversible causes, through study completion, an average of 15 months.
  Percentage of teams that correctly treat at least one reversible cause (hypovolemia or hypoglycemia).
Time to treatment of reversible causes from arrest recognition | Scenario will be video recorded and successively two independent video reviewers will assess the time to treatment of reversible causes, through study completion, an average of 15 months.
  Time from the recognition of cardiac arrest to the treatment of reversible causes, in seconds.
Time to treatment of reversible causes from the beginning of the scenario | Scenario will be video recorded and successively two independent video reviewers will assess the time to treatment of reversible causes, through study completion, an average of 15 months.
  Time from the beginning of the scenario to the treatment of reversible causes, in seconds.
Usability of the app - System Usability Scale | Questionnaires will be completed after each simulated scenario through study completion, an average of 15 months.
  To assess the PediAppRREST app usability, the team leaders of the intervention group will complete one validated questionnaire, the System Usability Scale (SUS). It consists of a 10-item questionnaire with five response options. Its scores ranges from a minimum of 0 to a maximum of 100. Higher scores corresponde to a better usability.
Usability of the app - Open-ended questions | Questionnaires will be completed after each simulated scenario through study completion, an average of 15 months.
  To further assess the PediAppRREST app usability, the team leaders of the intervention group will answer open-ended questions about app usability in a questionnaire.
Team leaders' workload | Questionnaires will be completed by team leaders after each simulated scenario through study completion, an average of 15 months.
  Team leaders' workload measured by the validated, multidimensional NASA-Task Load Index (NASA-TLX) questionnaire. The values of this score range from a minimum of 0 to a maximum of 100. A higher value means a higher perceived workload.
Cardiopulmonary resuscitation (CPR) quality - Mean chest compression rate | CPR quality data will be extracted by the manikin's software after each simulated scenario, through study completion, an average of 15 months.
  CPR quality will be measured by the Skill Reporter (Laerdal™), the software associated to the manikin (Resusci Junior, Laerdal™). Mean chest compression rate is expressed in number of compressions/minute.
Cardiopulmonary resuscitation (CPR) quality metrics - Mean chest compression depth | CPR quality data will be extracted by the manikin's software after each simulated scenario, through study completion, an average of 15 months.
  CPR quality will be measured by the Skill Reporter (Laerdal™), the software associated to the manikin (Resusci Junior, Laerdal™). The mean chest compression depth is reported in millimeters.
Cardiopulmonary resuscitation (CPR) quality metrics - Compression depth correctness | CPR quality data will be extracted by the manikin's software after each simulated scenario, through study completion, an average of 15 months.
  CPR quality will be measured by the Skill Reporter (Laerdal™), the software associated to the manikin (Resusci Junior, Laerdal™). Compression depth correctness is defined as the proportion of chest compressions with a correct depth of 50-60 mm, according to AHA standards.
Cardiopulmonary resuscitation (CPR) quality metrics - Chest compressions fraction | CPR quality data will be extracted by the manikin's software after each simulated scenario, through study completion, an average of 15 months.
  CPR quality will be measured by the Skill Reporter (Laerdal™), the software associated to the manikin (Resusci Junior, Laerdal™). The chest compression fraction is defined as the proportion of resuscitation time during which chest compressions are administered.
Team resuscitation performance | Scenario will be video recorded and successively evaluated by two independent video reviewers. Outcome assessors will score teams' performance by means of CPT using data extracted by video reviewers, through study completion, an average of 15 months.
  Team resuscitation performance will be evaluated using the Clinical Performance Tool (CPT). The CPT is a validated scoring system designed based on AHA PALS algorithms, through which sequence, timing, and quality of specific actions, during different simulated scenarios, can be assessed. Outcome assessors will use the CPT section for the asystole scenario to evaluate teams' performance. The values of this score range from a minimum of 0 to a maximum of 13. Higher scores correspond to a better team performance.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Bressan, MD, PhD, Principal Investigator — University of Padova; Francesco Corazza, MD, Principal Investigator — University of Padova
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Meyer, University of Firenze, Florence
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Università del Piemonte Orientale, Novara
  - Azienda Ospedale Università di Padova, University of Padova, Padua
  - Policlinico Universitario Agostino Gemelli, Università Cattolica del Sacro Cuore, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corazza F, Snijders D, Arpone M, Stritoni V, Martinolli F, Daverio M, Losi MG, Soldi L, Tesauri F, Da Dalt L, Bressan S. Development and Usability of a Novel Interactive Tablet App (PediAppRREST) to Support the Management of Pediatric Cardiac Arrest: Pilot High-Fidelity Simulation-Based Study. JMIR Mhealth Uhealth. 2020 Oct 1;8(10):e19070. doi: 10.2196/19070. PMID 32788142
- [Background] Wolfe HA, Morgan RW, Zhang B, Topjian AA, Fink EL, Berg RA, Nadkarni VM, Nishisaki A, Mensinger J, Sutton RM; American Heart Association's Get With the Guidelines-Resuscitation Investigator. Deviations from AHA guidelines during pediatric cardiopulmonary resuscitation are associated with decreased event survival. Resuscitation. 2020 Apr;149:89-99. doi: 10.1016/j.resuscitation.2020.01.035. Epub 2020 Feb 11. PMID 32057946
- [Derived] Corazza F, Arpone M, Tardini G, Stritoni V, Mormando G, Graziano A, Navalesi P, Fiorese E, Portalone S, De Luca M, Binotti M, Tortorolo L, Salvadei S, Nucci A, Monzani A, Genoni G, Bazo M, Cheng A, Frigo AC, Da Dalt L, Bressan S. Effectiveness of a Novel Tablet Application in Reducing Guideline Deviations During Pediatric Cardiac Arrest: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2327272. doi: 10.1001/jamanetworkopen.2023.27272. PMID 37535352
- [Derived] Corazza F, Arpone M, Snijders D, Cheng A, Stritoni V, Ingrassia PL, De Luca M, Tortorolo L, Frigo AC, Da Dalt L, Bressan S. PediAppRREST: effectiveness of an interactive cognitive support tablet app in reducing deviations from guidelines in the management of paediatric cardiac arrest: protocol for a simulation-based randomised controlled trial. BMJ Open. 2021 Jul 28;11(7):e047208. doi: 10.1136/bmjopen-2020-047208. PMID 34321297